CLINICAL TRIAL: NCT03068403
Title: Dynamic Contrast Enhanced Ultrasound for Predict and Assess Rectal Cancer Response After Neo-adjuvant Chemoradiation - RECT
Acronym: RECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2015/17
Record Dates: First submitted 2017-01-05; First posted 2017-03-01 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Rectal Cancer
Keywords: CEUS Perfusion; Rectal Cancer; Tumor Perfusion; Radiochemotherapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemotherapy and Radiochemotherapy (Other)
  Interventions: Procedure: Dynamic contrast enhanced ultrasound (D-CEUS) with Sonovue® administration
- Radiochemotherapy (Other)
  Interventions: Procedure: Dynamic contrast enhanced ultrasound (D-CEUS) with Sonovue® administration

INTERVENTIONS:
Procedure: Dynamic contrast enhanced ultrasound (D-CEUS) with Sonovue® administration — Dynamic contrast enhanced ultrasound (D-CEUS) with Sonovue® administration

SUMMARY:
In recent years the concept of organ sparing treatment in rectal cancer was introduced for selected good responders after neo-adjuvant treatment. In these patients replacement of the standard of care total mesorectal excision (TME) by transanal endoscopic microsurgery (TEM) or omission of surgery after chemoradiation (CRT) was proposed. Before organ sparing treatments could be applied in clinical practice a reliable patient selection procedure has to be available as only good treatment responders after neo-adjuvant therapy are candidates for such adapted therapy. Different imaging modalities have been studied for their ability to distinguish good treatment responders from others. Examples of such imaging modalities with some promising results regarding response assessment are fludeoxyglucosepositron emission tomography (FDG-PET), T2-weighted magnetic resonance imaging (T2w-MRI), dynamic contrast enhanced magnetic resonance imaging and diffusion weighted MR imaging (DW-MRI). Besides these modalities dynamic contrast enhanced ultrasound (D-CEUS) is a new modality used for tissue characterization and therapy response assessment in several tumor locations, like liver tumors and breast cancer. D-CEUS reflect tissue vascular perfusion. For rectal cancer, the value of D-CEUS for pathological response prediction and assessment has never been assessed. Therefore, in this study we assessed D-CEUS to predict and assess pathological response in rectal cancer after neo-adjuvant CRT.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed rectal carcinoma
* Stade ≥T2 and tumor size ≥3cm
* No detectable metastases
* Patient ≥ 18 years
* Patient information and written informed consent form signed
* Patient who can receive radiotherapy and chemotherapy
* Negative pregnancy test in women of childbearing potential
* Patient covered by a Social Security system

Exclusion Criteria:

* Indication for immediate surgery
* Primary tumor not measured at the MRI before inclusion
* Previous pelvic radiotherapy
* Contraindication to SONOVUE or MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2018-11-08 (Actual); Study Completion 2019-01-08 (Actual)

PRIMARY OUTCOMES:
Area under the echo-power curve (AUC) | At inclusion, 3 months and 6 months visits

SECONDARY OUTCOMES:
Peak enhancement (PE) | At inclusion, 3 months and 6 months visits
Rise time (RT) | At inclusion, 3 months and 6 months visits
Wash-in area under the curve (WiAUC) | At inclusion, 3 months and 6 months visits
Mean transit time (mTT) | At inclusion, 3 months and 6 months visits
Time to peak (TTP) | At inclusion, 3 months and 6 months visits
Whash-in rate (WiR) | At inclusion, 3 months and 6 months visits
Wash out rate (WoR) | At inclusion, 3 months and 6 months visits
MRI assessed Tumor Response Grade (mrTRG) | At inclusion, 3 months and 6 months visits
mrTNM staging | At inclusion, 3 months and 6 months visits

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud HOCQUELET, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No